CLINICAL TRIAL: NCT00627354
Title: Phase 2 Randomized Study Evaluating 3 Chemotherapy Regimens as Second-line Treatment in Patients With Hormone-refractory Metastatic Prostate Cancer
Brief Title: Mitoxantrone, Etoposide, and Vinorelbine As Second-Line Therapy in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe D'Etude des Tumeurs Uro-Genitales (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000574184; GETUG- P02; INCA-RECF0422; EUDRACT-2006-001597-25
Record Dates: First submitted 2008-02-29; First posted 2008-03-03 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2009-07

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Etoposide; Mitoxantrone; Prednisone; Vinorelbine

INTERVENTIONS:
Drug: etoposide
Drug: mitoxantrone hydrochloride
Drug: prednisone
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as mitoxantrone, etoposide, and vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known which drug is more effective in killing tumor cells.

PURPOSE: This randomized phase II trial is studying how well mitoxantrone works compared to etoposide or vinorelbine works as second-line therapy in treating patients with metastatic prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the palliative response rate in patients with hormone-resistant prostate cancer treated with mitoxantrone hydrochloride vs etoposide vs vinorelbine ditartrate as second-line therapy.

Secondary

* Determine the duration of palliative response in patients treated with these regimens.
* Determine the biological response (PSA > 50%) in these patients.
* Determine the time to progression (biological and clinical) in these patients.
* Determine the overall survival of these patients.
* Determine the quality of life and the impact on autonomy of patients over 70 years of age.
* Determine the toxicity of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive mitoxantrone hydrochloride IV over 5 minutes once a week for 3 weeks.
* Arm II: Patients receive oral etoposide twice daily on days 1-14.
* Arm III: Patients receive oral vinorelbine ditartrate once daily on days 1 and 8 and oral prednisone once daily on days 1-21.

Treatment in all three arms repeats every 3 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic progressive disease meeting the following criteria:

    * Increase in measurable lesions > 25%
    * Increase in bone lesions > 25%
    * Biological progression rate of PSA > 4 ng/mL
* Received docetaxel as first-line chemotherapy
* Received at least 1 prior regimen of hormone therapy
* Pain > 2 on Visual Analog Scale or continuing level 2 analgesics
* No symptomatic or evolutionary CNS disease

PATIENT CHARACTERISTICS:

* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times normal
* Alkaline phosphatase ≤ 2 times normal (unless bone metastases are present)
* Transaminases ≤ 1.5 times normal
* Bilirubin ≤ 1.5 times normal
* No prior malignancy except basal cell skin cancer
* No peripheral neuropathy or severe neuropathy ≥ grade 2
* No other severe lung, hepatic, renal, or digestive disease that would be complicated by treatment
* LVEF > 50%
* No history of peptic ulcer, unstable diabetes, or other contraindication to using steroids
* No severe infection requiring antibiotics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 8 weeks since prior metabolic radiotherapy
* More than 4 weeks since prior external radiotherapy
* At least 1 month since prior docetaxel-based chemotherapy
* At least 1 month since prior antiandrogen therapy in the case of complete hormonal blockage
* No participation in another clinical trial within the past 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-09; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Palliative response rate

SECONDARY OUTCOMES:
Duration of palliative response
Biological response
Tumor response as assessed by RECIST criteria
Time to progression
Overall survival
Quality of life as assessed by QLQ-PR25
Impact on autonomy in patients > 70 years of age
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Florence Joly, MD, PhD, Study Chair — Centre Francois Baclesse
Locations (1):
- Centre Regional Francois Baclesse, Caen, France